CLINICAL TRIAL: NCT03286439
Title: Recovery After Medical or Surgical Treatment - A Prospective Cohort Study
Brief Title: Recovery After Medical or Surgical Treatment
Status: Completed | Type: Observational
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Stine Estrup, Principal Investigator, Zealand University Hospital
Other Study IDs: NA-1-2017
Record Dates: First submitted 2017-09-14; First posted 2017-09-18 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Cognitive Deficit
MeSH Terms: conditions — Cognition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: there will be offered a follow up visit — The investigators will offer the patients a follow up visit 3 and 12 months after discharge from the hospital.

SUMMARY:
This study aims to investigate the in-hospital care as well as the cognitive status, quality of life, physical function and risk of anxiety and depression, sleep disorders and drug use in a Danish cohort of both medical and surgical patients with acute critical illness without admittance to ICU (Intensive Care Unit) treatment, at three and twelve months after hospital discharge.

DETAILED DESCRIPTION:
A stay at the ICU (intensive Care Unit) is related to life-threatening conditions and often displays a major impact on both physical and mental resources of the patients. Studies show that a great part of ICU patients have impairments of both physical and psychological kinds, some long-lasting. This condition is termed the "post intensive care syndrome" (PICS) and describes a wide range of symptoms as fatigue, depression, anxiety, memory loss along with both cognitive and physical impairments. Rehabilitative efforts are, thus, needed, and it has been suggested that ideally, rehabilitation should begin at the time of admission to the hospital and continue for a long time, possibly years, after the patient has been discharged. Regarding long term cognitive function of the ICU survivors in particular, recent studies have demonstrated severe impairment at the level of light Alzheimer's disease. In all of these studies, the reference group is the normal population, and it is a general problem that the cognitive and physical function of ICU patients before critical illness is unknown. There has recently been a norwegian study that included a reference group of surgical patients undergoing major surgery. The surgical group was older and more severely ill than the ICU group and was found to have a much worse cognitive function. Moreover, the cognitive function of the critically ill patients was not very far from the normal reference population due to selection.

To determine to which degree the impairments can be attributed to ICU-admission, the investigators need to look at a hospitalised and representative, non-ICU population, which is what will be done in the study. The investigators will therefore include patients that have been admitted to surgical or medical department acute without admittance to the ICU and contact these patients 3 and 12 months after admission. Where there will be performed different tests in order to evaluate the the cognitive status, quality of life, physical function and risk of anxiety and depression, sleep disorders and drug use.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years of age
* Admitted to surgical or medical department > 3 days
* Admitted with one of the following diagnoses:

  * Pneumonia
  * Heart failure
  * Pulmonary embolism
  * Acute myocardial infarction
  * Pyelonephritis
  * Patients undergoing non-elective open or laparoscopic abdominal surgery (not including elective procedures, diseases of the appendix, diseases of the gallbladder, liver, spleen, kidney, pancreas and emergency hernia surgery without bowel resection)

Exclusion Criteria:

* Permanently incompetent patients not able to consent
* Not able to speak and understand Danish
* Discharged from the hospital for terminal care
* Patients transferred to another hospital during the stay
* Patients living outside the Region of Zealand
* Patients admitted under duress or actively psychotic
* Patients that are blind or severely visually impaired.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of critically ill patients that have been admitted to surgical or Medical departement.
Sampling Method: Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2018-07-06 (Actual); Study Completion 2018-07-06 (Actual)

PRIMARY OUTCOMES:
Cognitive function | 3 months after discharge
  Cognitive Function measured by The Repeatable Battery for The Assesment of Neuropsychological Status (RBANS)

SECONDARY OUTCOMES:
Cognitive function after one year | 12 months after discharge
  Cognitive function measured with The Repeatable Battery for the Assessments of Neuropsychological Status (RBANS) evaluation at 12 months after discharge from hospital
Rehabilitation after 3 months | 3 months after discharge
  This will be investigated by filling out a checklist of community support and contact to health care system at 3 month follow up
Self-reported health related quality of life | 3 months after discharge
  This will be investigated by filling out a questionnaire named SF 36, Short Form Health Survey.
Self-reported health related quality of life | 12 months after discharge
  This will be investigated by filling out a questionnaire named SF 36, Short Form Health Survey.
Objective assessment of physical function | 3 months after discharge
  This will be investigated by filling out a checklist called CPAx, The Chelsea Critical Care Physical Assessment Tool.
Objective assessment of physical function | 12 months after discharge
  This will be investigated by filling out a checklist called CPAx, The Chelsea Critical Care Physical Assessment Tool
Mortality | 90 days after discharge
  The mortality of the patients within 90 days after hospital discharge.
Consumption of opioids | 90 days after discharge
  Percentage of patients with a daily consumption of opioids at hospital admission and 90 days after discharge
Consumption of statins days after discharge | 90 days after discharge
  Percentage of patients with a daily consumption of statins at hospital admission and at 90 days after discharge
Consumption of anti-depressants | 90 days after discharge
  Percentage of patients with a daily consumption of anti-depressants at hospital admission and at 90 days after discharge
Sleepiness | At inclusion
  This will be investigated by filling out Epworth Sleepiness Scale
Sleepiness | 3 months after discharge
  This will be investigated by filling out Epworth Sleepiness Scale
Sleepiness | 12 months after discharge
  This will be investigated by filling out Epworth Sleepiness Scale
Insomnia | At inclusion
  This will be investigated by filling out Insomnia Severity Index
Insomnia | 3 months after discharge
  This will be investigated by filling out Insomnia Severity Index
Insomnia | 12 months after discharge
  This will be investigated by filling out Insomnia Severity Index
Sleep Quality | At inclusion
  This will be investigated by filling out Pittsburgh Sleep Quality Index
Sleep Quality | 3 months after discharge
  This will be investigated by filling out Pittsburgh Sleep Quality Index
Sleep Quality | 12 months after discharge
  This will be investigated by filling out Pittsburgh Sleep Quality Index
Information processing speed | 3 months after discharge
  This will be investigated by filling out the Trail Making Test Part A
Information processing speed | 12 months after discharge
  This will be investigated by filling out the Trail Making Test Part A
Executive function | 3 months after discharge
  This will be investigated by filling out the Trail Making Test Part B
Executive function | 12 months after discharge
  This will be investigated by filling out the Trail Making Test Part B
Rehabilitation after 12 months | 12 months
  This will be investigated by filling out a checklist of Community support and contact to health care system at 3 month follow up
Consumption of sleep medication | At inclusion
  Percentage of patients with a daily consumption of sleep medication at hospital admission and 90 days after discharge
Consumption of sleep medication | 90 days after discharge
  Percentage of patients with a daily consumption of sleep medication at hospital admission and 90 days after discharge
Consumption of sleep medication | 12 months after discharge
  Percentage of patients with a daily consumption of sleep medication at hospital admission and 90 days after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Stine Estrup, MD, Principal Investigator — Stine Estrup
Locations (1):
- Zealand University Hospital, Køge, Denmark

IPD SHARING:
Plan to Share IPD: No